CLINICAL TRIAL: NCT06326827
Title: Study of the Osteoconductive Potential of the Injectable Bone Substitute In'Oss™ (MBCP® Putty) in the Filling of Orthopaedic Bone Defects
Brief Title: In'Oss™ (MBCP® Putty) Ortho
Status: Not yet recruiting | Type: Observational
Sponsor: Advanced Medical Solutions Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: P231127IBSORTHO
Record Dates: First submitted 2024-03-18; First posted 2024-03-22 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-02

CONDITIONS: Orthopedic Disorder; Trauma Injury; Extremity Injury
Keywords: Proximal humerus; Distal radius; Distal femur; Proximal tibia; Distal tibia; Fracture; MBCP Putty; Bone defect reconstruction
MeSH Terms: conditions — Musculoskeletal Diseases; Accidental Injuries; Fractures, Bone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- In'Oss™ (MBCP® Putty): Participants will be recruited from a population who are undergoing orthopaedic bone trauma surgery at the investigational site. All admitted patients will be screened and assessed to determine whether patients may be eligible to take part based on the inclusion and exclusion criteria. Patient participation in this study will include a screening visit within 48 hours of admission to hospital prior the surgery.
  Interventions: Device: In'Oss™ (MBCP® Putty)

INTERVENTIONS:
Device: In'Oss™ (MBCP® Putty) — Use of In'Oss™ (MBCP® Putty) in surgical procedure to correct epiphyso-metaphyseal and/or metaphyso-diaphyseal bone defect in one of the following anatomical locations: Proximal humerus, Distal radius, Distal femur, Proximal tibia, Distal tibia.

SUMMARY:
Study of the osteoconductive potential of the injectable bone substitute In'Oss™ (MBCP® Putty) in the filling of orthopaedic bone defects to collect Post-Market Clinical Follow-up (PMCF) data for the CE-marked In'Oss™ (MBCP® Putty) device in the orthopaedic trauma surgery

DETAILED DESCRIPTION:
The In'Oss™ (MBCP® Putty) device is an Injectable Bone Substitute (IBS) whose purpose is a bone gap and void filler. It forms a putty-like synthetic bone graft which molds to the shape of the defect. It is composed of Hydroxyapatite (HA), Beta Tricalcium Phosphate (ß-TCP) and a hydrogel and is presented in sterile syringes.

The Injectable Bone Substitute In'Oss™ is intended for use to reconstruct bony voids or bone gaps of the skeletal system (e.g. extremities, spine and pelvis). The performances of the Injectable Bone Substitute In'Oss™ (MBCP® Putty) are the filling of bone defects and the bony ingrowth from local osseous tissue onto the surface of the product (osteoconduction process).

The purpose of this study is primarily to collect Post-Market Clinical Follow-up (PMCF) data on the performance and safety of the CE marked In'Oss™ device in the orthopaedic application. The data and conclusions obtained from this study by the Sponsor Advanced Medical Solutions Ltd. (AMS) together with the manufacturer Biomatlante will be used to provide clinical evidence for the clinical evaluation process.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is male or female, 18 - 85 years old;
2. Patient is willing and able to give written informed consent;
3. Patient is able to comply with a prior medical examination;
4. Patient is or has been scheduled for a surgical procedure to correct epiphyso-metaphyseal and/or metaphyso-diaphyseal bone defect in one of the following anatomical locations:

   * Proximal humerus ▪ Distal radius
   * Distal femur ▪ Proximal tibia ▪ Distal tibia
5. Patient is willing and able to comply with the study procedures during surgery and the post-surgical follow up period, up to 12 months.

Exclusion Criteria:

1. Patient has had an infection in the same extremity within last 24 months;
2. Patient has signs of necrosis at the surgical site;
3. Patient has cellulitis;
4. Patient has granuloma or non-curetted cyst;
5. Patient has an history of uncontrolled diabetes;
6. Patient is alcoholic and/or heavy smoker (> 20 cigarettes per day);
7. Patient has a congenital or acquired immunodeficiency;
8. Patient has severe bone loss (≥ 40cm3);
9. Patient is on long-term steroidal therapy or treatment acting on the calcium or phosphorus metabolism;
10. Patient is or has been scheduled for surgery that would involve intra-articular implantation of the study device;
11. Patient who has or had an uncontained bone defect created as a result of trauma injury or surgically created;
12. Patient was exposed to any radiation (e.g. X-Rays, handling of radiolabelled materials) other than the normal background radiation within the 12 months before the screening visit;
13. Patient is pregnant;
14. Patient who is an employee at the study site;
15. Patient is known to be non-compliant with medical treatment or follow-up
16. Patient has any significant or unstable medical/psychiatric condition that, in the opinion of the Investigator, would interfere with their ability to participate in the study;
17. Patient is currently enrolled or planning to enrol in another clinical study or treatment with another investigational drug/device that may interfere with the assessments, visits or outcomes of this study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study aims to include 100 adult patients male and female to be enrolled in this study. The sample size is based on formal calculations to demonstrate effectiveness (see section 10 for detail). The Sponsor expects to enrol 100% of the patients at one (1) investigational site in the UK.
  All adults aged between 18 to 85 years old will be screened for the study. If the patients meet all inclusion criteria, but none of the exclusion criteria, the patients will be asked to participate in this study.
  Prior to enrolment in this study, all patients will undergo a general medical evaluation to assess co-morbidities, and risk factors associated with their disease. All patients must be fit for anaesthetic and surgery.
  In cases where it is not possible for subjects to provide written informed consent prior to surgery, screening (Visit 1) assessments will be performed as soon as possible after surgery (no later than 48 hours after surgery), after written informed consent has been obtained.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Successful bone defect reconstruction in the extremities | At 12 months post-surgery
  Evaluation of performance of the In'Oss™ (MBCP® Putty) through the achievement of successful bone fusion through radiological evaluation (X-Ray) within 12 months by assessing interdigitation in 3 out of 4 planes (anterior/posterior/lateral/medial).

SECONDARY OUTCOMES:
Evaluation of functional mobility restoration in the upper limb with PRO measures | Within 12 months post-surgery
  Functional mobility restoration in the upper limb after use of In'Oss™ (MBCP® Putty) in bone defect reconstruction by scoring patient's physical disability and symptoms through patient-reported outcome measure (Quick Disabilities of the Arm, Shoulder and Hand (QuickDASH)
Evaluation of functional mobility restoration in the lower limb with PRO measure | Within 12 months post-surgery
  Functional mobility restoration in the lower limb after use of In'Oss™ (MBCP® Putty) in bone defect reconstruction by scoring patient's physical disability and symptoms through patient-reported outcome measure: Lower Extremity Functional Scale (LEFS)
Evaluation of patient's pain intensity with VAS pain scale | Within 12 months post-surgery
  Patient's pain intensity at trauma/surgical site evaluated with Visual Analog Scale (VAS) pain scale after use of In'Oss™ (MBCP® Putty) in bone defect reconstruction in the extremities.
  0 = no pain; 10 = worst pain imagineable.
Evaluation of safety of In'Oss | Within 12 months post-surgery
  Incidence of device related Adverse Events after use of In'Oss™ (MBCP® Putty) in bone defect reconstruction in the extremities.
Evaluation of device usability | Within 12 months post-surgery
  Clinician satisfaction with use of In'Oss™ (MBCP® Putty) as per Instructions for Use (IFU) in bone defect reconstruction in the extremities.
  0 = very unsatisfied; 5 = very satisfied.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Giannoudis, Principal Investigator — Leeds General Infirmary, Great George Street Leeds LS1 3EX, United Kingdom

IPD SHARING:
Plan to Share IPD: No